CLINICAL TRIAL: NCT03460834
Title: Obesity and Asthma: Unveiling Metabolic and Behavioral Pathways
Brief Title: Asthma and Obesity: Observational
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of Colorado, Denver (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Juan P Wisnivesky, Professor of Medicine and Chief, Division of General Internal Medicine, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 14-1859 O; R01HL129198 (NIH)
Record Dates: First submitted 2018-03-02; First posted 2018-03-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Asthma; Obesity
Keywords: Asthma; Obesity; Observational Study
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obese asthmatic patients: Observational Cohort

SUMMARY:
Obesity is associated with poor asthma control and greater healthcare utilization and costs. In this study the researchers will examine the biologic and behavioral interrelationships between these conditions and their impact on outcomes. Towards this end, the researchers will conduct an observational prospective cohort study of 400 obese asthmatic patients treated at institutions in New York City and Denver, and develop and pilot test educational and counseling modules that take an integrated approach to asthma and obesity self-management support.

DETAILED DESCRIPTION:
The objective of this study is to examine novel biological and behavioral pathways that may explain the association of obesity with asthma morbidity, and develop and pilot test educational and counseling modules, based on self-regulation theory, that take an integrated approach to asthma and obesity self-management support.

The Specific Aims are to:

1. Compare the longitudinal relationship between L-arginine/ADMA balance and morbidity (lung function, asthma control, acute resource utilization, and quality of life) between obese adults with late onset asthma vs. (a) obese adults with early onset asthma and non-obese asthmatics with early (b) or late (c) onset disease. Age of asthma onset is as categorized as early when developed ≤12 years of age or late when developed >12 years of age.
2. Evaluate the interrelationship between obesity- and asthma-related illness beliefs, and the impact of cognitive function, on patients' management of these conditions over time

ELIGIBILITY:
Inclusion Criteria:

* >21 years with a diagnosis of asthma made by a health care provider and evidence of airway reactivity (increase in FEV1 >12% and >200 ml after bronchodilators or positive methacholine test) in prior lung function testing or baseline spirometry;
* prescribed an asthma controller medication;
* English or Spanish speaking.

Exclusion Criteria:

* chronic obstructive lung disease (COPD) or other chronic respiratory illness; - >15 pack-year smoking history because of the possibility of undiagnosed COPD;
* diagnosis of dementia identified in the clinical record.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A description of the population from which the groups or cohorts will be selected (for example, primary care clinic, community sample, residents of a certain town).
Sampling Method: Non-Probability Sample
Enrollment: 333 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume (FEV1) | 18 months
  Forced expiratory volume (FEV1) measures how much air a person can exhale during the first second of a forced breath, performed by spirometry.
Exhaled Nitric Oxide (eNO) | 18 months
  eNO is the most widely used and standardized noninvasive biomarker that evaluates airway inflammation in asthma. measured before spirometry using the NIOX MINO system (Aerocrine AB, Stockholm, Sweden) following established procedures. Current guidelines do not yet specify ''normal'' values; however, eNO levels >20-25ppb have been used as cut-points indicating airway inflammation and the need to change treatment.
Asthma Control Questionnaire (ACQ) | 18 months
  The ACQ has 7 items: 5 items-self administered for symptoms, 1 item self administered rescue inbronchodilator use, and 1 item FEV1% completed by provider. 7-point scale from 0 = no impairment to 6 = maximum impairment. The questions are equally weighted and the ACQ score is the mean of the 7 questions, with total score range between 0 (totally controlled) and 6 (severely uncontrolled).

SECONDARY OUTCOMES:
Asthma Controller Medication Adherence | 4 weeks
  objectively measure ICS adherence using the Smartinhaler (Nexus6, Franklin, OH) or Doser electronic devices (Meditrack, MA) for metered dose inhalers (MDIs) and the Smartdisk (Nexus6, Franklin, OH) for dry powder inhalers (DPIs) for 4 weeks after each in-person interview. Adherence will be defined as use of medications on ≥80% of days prescribed, a commonly applied convention.
The Medication Adherence Rating Scale (MARS) | 18 months
  A 10-item self-reported questionnaire resulting from the combination of the Medication Adherence Questionnaire and the Drug Attitude Inventory. The MARS contains 10 yes/no item and the sum of items yields a final score ranking from 0 (poor adherence to treatment) to 10 (good adherence to treatment).
Food Behavior Checklist | 18 months
  16 question survey. Each question represents a certain value (1 - 4) that when added collectively predicts the quality of person's food consumption habits. The higher the score, the more optimal the habits.
Physical activity level | 18 months
  Physical activity: levels will be assessed using an ActiGraph wGT3X-BL triaxial accelerometer (ActiGraph LLC; Pensacola, FL) worn on the waist for 7 days after each in person visit. The ActiGraph has been validated for physical activity and sedentary time in laboratory and field settings. Data from the monitor will be output as activity counts then converted to step counts and time spent in different intensities of activity using previously determined cut-points.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P. Wisnivesky, MD, DrPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Alex D. Federman, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Fernando Holguin, MD, MPH, Principal Investigator — University of Colorado Denver, Anschutz Medical Campus
Locations (2):
- United States (2):
  - University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided